CLINICAL TRIAL: NCT03168841
Title: Efficacy and Safety of Efinaconazole 10% Solution in the Treatment of Onychomycosis in Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-26
Record Dates: First submitted 2017-05-11; First posted 2017-05-30 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — efinaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Group, receiving medication (Experimental): Enrolled subjects with confirmed onychomycosis will be dispensed topical medication for treatment.
  Interventions: Drug: Efinaconazole Topical

INTERVENTIONS:
Drug: Efinaconazole Topical — Enrolled subjects will be dispensed medical for topical application, and followed for a period of 50 weeks.

SUMMARY:
Onychomycosis, a common pathology of the toenails, is even more prevalent among diabetic subjects. Nearly 26 million Americans suffer from diabetes, and approximately one-third of subjects with diabetes have toenail onychomycosis. Numerous studies have addressed the efficacy and safety of both topical and oral antifungal treatment options for onychomycosis in diabetic subjects. However, no study to date has specifically addressed the efficacy and safety of efinaconazole among diabetic subjects.

The objective of this noncomparative, uncontrolled study is to determine the efficacy of topical efinaconazole 10% for toenail onychomycosis among subjects with diabetes mellitus. Specific indicators to measure efficacy of treatment will be the mycological cure rate, complete cure rate, and treatment success. Furthermore, an additional goal of the study is to gain knowledge of safety in the setting of a cohort of diabetic subjects

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of onychomycosis confirmed through positive KOH stain or positive mycologic culture findings.
* Involvement of at minimum 20% of the target great toenail.

Exclusion Criteria:

* Diagnosis of a nondermatophyte fungus infection, diagnosis of proximal subungual onychomycosis, diagnosis of superficial white onychomycosis
* Diagnosis of peripheral arterial disease or anatomic abnormalities of the target toenail
* Inability to follow through with all requisite office visits
* Routine use of a systemic corticosteroid, routine use of a systemic immunomodulator, or history of systemic antifungals within the prior five years.
* Active interdigital tinea pedis refractory to topical antifungal treatments
* Known hypersensitivity to efinaconazole
* Use, within the month preceding screening, of: topical antifungal agents, topical anti-inflammatory agents to the toes
* Any history of oral systemic antifungal with known activity against dermatophytes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group, Receiving Medication
Started | 40
Completed | 36
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.15 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic | 31
  Race/Ethnicity: African-American | 4
  Race/Ethnicity: White | 4
  Race/Ethnicity: Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint - Efficacy
Description: The primary efficacy end point is the proportion of subjects achieving complete cure at week 50. Complete cure is to be defined as a combination of 0% clinical involvement and mycological cure (mycological cure defined as negative KOH examination and negative fungal culture of the target toenail sample).
Time Frame: 50 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 36
Participants | 4

2. Secondary Outcome: Secondary Endpoint - Efficacy
Description: The first secondary efficacy end point is mycological cure, defined as negative KOH examination and negative fungal culture of the target toenail sample.
Time Frame: 50 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 36
Participants | 21

3. Secondary Outcome: Secondary Endpoint - Efficacy
Description: The second secondary efficacy end point is clinical cure, defined as 0% clinical involvement of the target toenail.
Time Frame: 50 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 40
Participants | 8

4. Secondary Outcome: Secondary Endpoint - Safety (Occurrence of Adverse Events: Type and Frequency)
Description: The secondary safety endpoint is the occurrence of adverse events (type and frequency).
Time Frame: 50 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group, Receiving Medication
Number analyzed (Participants) | 40
Participants | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Group, Receiving Medication
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group, Receiving Medication (N=40)
Application site vesicles, local (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT03168841/Prot_SAP_000.pdf